CLINICAL TRIAL: NCT00957203
Title: Long-Term Safety Study of KW-6002 (Istradefylline) in the Treatment of Parkinson's Disease (Phase 3)
Brief Title: Long-Term Safety Study of KW-6002 (Istradefylline) in Parkinson's Disease Patients
Acronym: 6002-010
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6002-010
Record Dates: First submitted 2009-08-07; First posted 2009-08-12 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Istradefylline (Experimental)
  Interventions: Drug: Istradefylline

INTERVENTIONS:
Drug: Istradefylline — Oral istradefylline (KW-6002) 20 or 40 mg once daily
  Other Names: KW-6002

SUMMARY:
Patients with Parkinson's disease who completed the prior double-blind study 6002-009 are eligible to enter into this long-term study. The purpose of this study is to evaluate the safety and efficacy of KW-6002 administered long-term in patients with advanced Parkinson's disease treated with levodopa.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to give written informed consent
2. Completion of the study 6002-009

Exclusion Criteria:

1. Mini-mental status examination score of 23 or less
2. Less than 70% of compliance in the study 6002-009
3. Emergency deviation in the study 6002-009
4. Pregnant females

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adverse events

SECONDARY OUTCOMES:
Reducing the mean total hours of awake time per day spent in the OFF state
Reducing the mean percentage of awake time per day spent in the OFF state
Mean change in the total hours and the percentage of awake time per day spent in the ON state (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia)
Change in Unified Parkinson's Disease Rating Scale (UPDRS)
Change in the Clinical Global Impression - Improvement scale (CGI-I)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Tokyo, Japan